CLINICAL TRIAL: NCT05855577
Title: -Clinical Efficacy of Pharmacological Treatments Targeting Energy Metabolism, Evaluated by Gait Analysis, on Motor Function in Parkinson's Disease Patients
Brief Title: Motor Function Efficacy of Pharmacological Treatments Targeting Energy Metabolism, in Parkinson's Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: Università Foro Italico Roma (Other); CNR Pisa (Unknown)
Responsible Party: Principal Investigator, Antonella Peppe, MD, PhD, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RF-2021-12374979
Record Dates: First submitted 2023-02-28; First posted 2023-05-11 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Gait Analysis; Therapy, Directly Observed; Metabolic Disease
Keywords: parkinson's disease; gait Analysis; mitocondrial; therapy
MeSH Terms: conditions — Parkinson Disease; Directly Observed Therapy; Metabolic Diseases | interventions — Terazosin; Lisosan G

STUDY DESIGN:
Intervention Model Description: 25 M-PD (H&Y< 2.5) and 25 S-PD (H&Y > 2.5) patients with idiopathic PD will be enrolled sequentially in the randomized double-blind, double-dummy study.
Who Masked: Participant, Investigator
Masking Description: The investigators that visit the patient and perform Gait Analysis are Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Terazosine (Experimental): Pharmacological Treatment of Pakinson's disease patients using Terazosin 2 mg
  Interventions: Drug: Terazosin
- placebo T (Placebo Comparator): Pharmacological Treatment of Parkinson's disease patients using Placebo
  Interventions: Drug: Terazosin
- Lisosan-G (Nutritional Supplement) (Experimental): Treatment of Parkinson's disease patients using Lisosan-G
  Interventions: Drug: Terazosin
- Lisosan_G Placebo (Placebo Comparator): Treatment of Parkinson's disease patients using Lisosan-G
  Interventions: Drug: Terazosin

INTERVENTIONS:
Drug: Terazosin — Treatment of Terazosine vs placebo and Lisosan-G vs placebo in cross-over double-blind, double-dummy
  Other Names: Lisosan-g

SUMMARY:
Consistent evidence suggests that mitochondrial dysfunction plays a crucial role in Parkinson¿s disease pathogenesis.

Inhibition of complex I of the mitochondrial electron transport chain is sufficient to reproduce biochemical and pathological features of Parkinson¿s Disease in animal models (PD). Alterations of mitochondrial energy metabolism may intervene in PD pathogenesis by inducing inflammation, generation of reactive oxygen species (ROS), and neurodegeneration. The Nuclear factor erythroid 2-related factor 2 (Nrf2) is a regulator both of mitochondrial function and biogenesis, and of cellular resistance to oxidative stress, and may represent a novel target of PD disease-modifying therapies.

The aims of the present study are to validate indicators of energy metabolism as biomarkers in PD patients and to evaluate the efficacy of drugs and natural food supplements acting on the Nrf2 pathway in improving motor impairment and Gait in PD patients.

DETAILED DESCRIPTION:
Bradykinesia, causing impairment of gait and an associated significant risk of falls, is among the most debilitating core features of Parkinson¿s disease (PD), a movement disorder characterized by the degeneration of Substantia nigra dopaminergic neurons. The pacemaking action potential firing activity of nigral neurons requires high energy consumption and is coupled to large cytosolic calcium oscillations, which influence mitochondrial respiration, energy metabolism, and reactive oxygen species (ROS) production. Mitochondrial dysfunction, on the other hand, can drive dysregulation of calcium homeostasis, especially in dopaminergic neurons, and is recognized as a key component in PD progression. Notably, both calcium-binding and increased ROS production, resulting from inefficiencies in the mitochondrial electron transport chain, can trigger alpha-synuclein aggregation, thus contributing to neuronal loss and disease progression in PD. The Nuclear factor erythroid 2- related factor 2 (Nrf2) is a regulator of mitochondrial function and biogenesis, and cellular resistance to oxidative stress. Bioactive compounds activating the Nrf2 signaling pathway ameliorate Parkinsonian phenotypes in experimental models, suggesting the Nrf2 pathway potential novel therapeutic target in PD.

Bradykinesia, causing impairment of gait and an associated significant risk of falls, is among the most debilitating core features of PD. PD gait is characterized by shuffling steps accompanied by a stooped posture. In advanced PD, other complications may arise such as disturbances in speech, gait, posture, and balance, as well as hypomimia, impaired decision-making, alertness, and regulation of emotions.

The increased energy demand associated with bradykinesia is coupled with the impairment of energy metabolism in Parkinsonians, negatively affecting walking, gait, and postural stability, suggesting that the modulation of mitochondrial energy metabolism may ameliorate gait and postural stability in Parkinsonians. Cardinal symptoms of PD: Tremors, Rigidity, Bradykinesia, and postural instability, all elements that lead in almost all patients to a walking disorder. In fact, walking in Parkinson's disease is present since in the early stages of the disease, the step is reduced in length and speed, the swinging phase of the step (swing) is reduced, while the support (Stance) single and double is increased in duration. Progression as well as the severity of disease over time, leads to a significant increase in the risk of falls, inducing a reduction in autonomy in daily living activity. As mentioned Gait is influenced in a principal way. Bipedal walking, in humans, is well orchestrated, consistent with the intrinsic "kinetic melody". This "melody" in subjects with PD is altered appears clear that the analysis of the gait represents a key element for establishing functional recovery therapies aimed at restoring motor skills. Therefore, it seems sensible to hypothesize that energy metabolism parameters may represent reliable biomarkers in PD and that the Nrf2 pathway may be a new therapeutic target for the recovery of motor function in PD patients. Not only that, but the identification of reliable biomarkers that are easy to measure over time can aid in the diagnosis, and possible prognosis, and improve management.

In support of this view, PD pathogenesis is known to involve the loss of the homeostatic functions controlling mitochondrial energy metabolism. The transcription factor Nrf2 is a master controller of these functions. Notably, Nrf2 activity is compromised during aging and in neurodegenerative diseases.

The investigators hypothesize that energy metabolism parameters may represent reliable biomarkers in PD and that the Nrf2 pathway may be a novel therapeutic target for the rescue of motor function in Parkinsonians.

The identification of reliable biomarkers, easy to measure over time, is fundamental to facilitating diagnosis, prognosis, and better management of PD patients. The proposed study on PD patients will provide information immediately transferable to the clinical practice. Additionally, the clinical trial planned in the present project will provide substantial information regarding the effectiveness of different pharmacological approaches targeting the Nrf2 pathway in ameliorating gait and balance in Parkinsonians, thus reducing the substantial social and economic burden of PD to society, patients, and caregivers. Many drugs and natural food supplements acting on the Nrf2 pathway are available; therefore, the transfer to the clinical practice of the results of the present project is expected to be rapid.

ELIGIBILITY:
Inclusion Criteria:

* Patient with rigid-acinetic bilateral PD form
* At least 5 years of disease history
* H&Y between 2-3.5
* Stable drug therapy response without any change performed in the 3 months before the study.
* MMSE>24/30 (Mini-Mental State Examination)
* No severe gastrointestinal pathologies.

Exclusion Criteria:

* Systemic illness
* Presence of cardiac pacemaker
* Presence of deep brain stimulation
* Presence of severe dysautonomia with marked hypotension
* Obsessive-Compulsive Disorder (OCD)
* Major depression
* Dementia
* History or active neoplasia
* Pregnancy
* Lack of autonomy in walking;
* Malabsorption and gastrointestinal disorders;
* Gluten intolerance
* Ipotiroidism

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation, Gait Analysis and Metabolic variables efficacy of therapy | 2year
  MD UPDRs : Four Parts: II questionary by Parkinsonian or care-given, III-IV: Motor Part and Complication by neurologist , Each item rate from 0: no sign to 4: max sign PDQ39 questionary performed by Parkinsonian each item rate from 0: never, to 5:always. Gait Analysis following spatio-temporal parameters will be taken in to account: Right and Left Step Length, Stride time% Stance Swing , Double support t, Mean Velocity, Cadence, Stepwidth, and t for turning task:• Number of steps to complete the lap,• Lap time, Metabolomic Variables: Steady State oxygen uptake (VO2, mlkg-1min-1) and carbon dioxide production (VCO2), heart rate (HR), Walking energy cost per unit of time-WECt8Jkg-1min-1),Metabolic human blood variabes : G6PD mU/109 erytrocytes, CAT, GPx, NQO1,HO-1,SOD: U/mg protein, GSH mmol GSH/l, MDA mmol/MDA/l,NrF2 gene expression

SECONDARY OUTCOMES:
The efficacy and molecular mechanisms of Nrf2 pathway modulation in PD rodent models | 2 years
  Animal models allow an in-depth analysis, in strictly controlled experimental conditions, of several biological parameters, both at the peripheral level and in the brain, in relation to the expression of a motor phenotype. First, protein levels and mRNA expression of markers of energy metabolism will be measured both in the blood and in relevant brain areas of a group of PD and control rodents..
  Electrophysiological recordings and intracellular calcium measurements from striatum and substantia nigra neurons in acute slices of PD and control rodents will allow an analysis of the correlation between the biomarker profile, the neuronal function, and the parkinsonian motor behavior. In a second phase, we will test the efficacy of in vivo treatments with different modulators of the Nrf2 pathway in rescuing the PD model¿s motor behavior, energy metabolism biomarkers, and both striatal and substantia nigra neuron physiology.
  See metabolic human blood variables

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Peppe, MD, PhD, Principal Investigator — IRCCS Fondazione Santa Lucia Roma-Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amato R, Rossino MG, Cammalleri M, Timperio AM, Fanelli G, Dal Monte M, Pucci L, Casini G. The Potential of Lisosan G as a Possible Treatment for Glaucoma. Front Pharmacol. 2021 Jul 28;12:719951. doi: 10.3389/fphar.2021.719951. eCollection 2021. PMID 34393798
- [Background] Barichella M, Cereda E, Pinelli G, Iorio L, Caroli D, Masiero I, Ferri V, Cassani E, Bolliri C, Caronni S, Maggio M, Ortelli P, Ferrazzoli D, Maras A, Riboldazzi G, Frazzitta G, Pezzoli G. Muscle-targeted nutritional support for rehabilitation in patients with parkinsonian syndrome. Neurology. 2019 Jul 30;93(5):e485-e496. doi: 10.1212/WNL.0000000000007858. Epub 2019 Jul 5. PMID 31278117
- [Background] Belluscio V, Iosa M, Vannozzi G, Paravati S, Peppe A. Auditory Cue Based on the Golden Ratio Can Improve Gait Patterns in People with Parkinson's Disease. Sensors (Basel). 2021 Jan 29;21(3):911. doi: 10.3390/s21030911. PMID 33573043
- [Background] Bonsi P, Ponterio G, Vanni V, Tassone A, Sciamanna G, Migliarini S, Martella G, Meringolo M, Dehay B, Doudnikoff E, Zachariou V, Goodchild RE, Mercuri NB, D'Amelio M, Pasqualetti M, Bezard E, Pisani A. RGS9-2 rescues dopamine D2 receptor levels and signaling in DYT1 dystonia mouse models. EMBO Mol Med. 2019 Jan;11(1):e9283. doi: 10.15252/emmm.201809283. PMID 30552094
- [Background] Christiansen CL, Schenkman ML, McFann K, Wolfe P, Kohrt WM. Walking economy in people with Parkinson's disease. Mov Disord. 2009 Jul 30;24(10):1481-7. doi: 10.1002/mds.22621. PMID 19441128
- [Background] Cuadrado A. Brain-Protective Mechanisms of Transcription Factor NRF2: Toward a Common Strategy for Neurodegenerative Diseases. Annu Rev Pharmacol Toxicol. 2022 Jan 6;62:255-277. doi: 10.1146/annurev-pharmtox-052220-103416. Epub 2021 Oct 12. PMID 34637322
- [Background] Giordano N, Iemolo A, Mancini M, Cacace F, De Risi M, Latagliata EC, Ghiglieri V, Bellenchi GC, Puglisi-Allegra S, Calabresi P, Picconi B, De Leonibus E. Motor learning and metaplasticity in striatal neurons: relevance for Parkinson's disease. Brain. 2018 Feb 1;141(2):505-520. doi: 10.1093/brain/awx351. PMID 29281030
- [Background] Gruetter R, Tkac I. Field mapping without reference scan using asymmetric echo-planar techniques. Magn Reson Med. 2000 Feb;43(2):319-23. doi: 10.1002/(sici)1522-2594(200002)43:23.0.co;2-1. PMID 10680699
- [Background] Guatteo E, Yee A, McKearney J, Cucchiaroni ML, Armogida M, Berretta N, Mercuri NB, Lipski J. Dual effects of L-DOPA on nigral dopaminergic neurons. Exp Neurol. 2013 Sep;247:582-94. doi: 10.1016/j.expneurol.2013.02.009. Epub 2013 Feb 26. PMID 23481547
- [Background] Guatteo E, Rizzo FR, Federici M, Cordella A, Ledonne A, Latini L, Nobili A, Viscomi MT, Biamonte F, Landrock KK, Martini A, Aversa D, Schepisi C, D'Amelio M, Berretta N, Mercuri NB. Functional alterations of the dopaminergic and glutamatergic systems in spontaneous alpha-synuclein overexpressing rats. Exp Neurol. 2017 Jan;287(Pt 1):21-33. doi: 10.1016/j.expneurol.2016.10.009. Epub 2016 Oct 20. PMID 27771352
- [Background] Heger LM, Wise RM, Hees JT, Harbauer AB, Burbulla LF. Mitochondrial Phenotypes in Parkinson's Diseases-A Focus on Human iPSC-Derived Dopaminergic Neurons. Cells. 2021 Dec 7;10(12):3436. doi: 10.3390/cells10123436. PMID 34943944
- [Background] Imbriani P, Tassone A, Meringolo M, Ponterio G, Madeo G, Pisani A, Bonsi P, Martella G. Loss of Non-Apoptotic Role of Caspase-3 in the PINK1 Mouse Model of Parkinson's Disease. Int J Mol Sci. 2019 Jul 11;20(14):3407. doi: 10.3390/ijms20143407. PMID 31336695
- [Background] Imbriani P, D'Angelo V, Platania P, Di Lazzaro G, Scalise S, Salimei C, El Atiallah I, Colona VL, Mercuri NB, Bonsi P, Pisani A, Schirinzi T, Martella G. Ischemic injury precipitates neuronal vulnerability in Parkinson's disease: Insights from PINK1 mouse model study and clinical retrospective data. Parkinsonism Relat Disord. 2020 May;74:57-63. doi: 10.1016/j.parkreldis.2020.04.004. Epub 2020 Apr 20. PMID 32335490
- [Background] Iosa M, Morone G, Fusco A, Marchetti F, Caltagirone C, Paolucci S, Peppe A. Loss of fractal gait harmony in Parkinson's Disease. Clin Neurophysiol. 2016 Feb;127(2):1540-1546. doi: 10.1016/j.clinph.2015.11.016. Epub 2015 Dec 2. PMID 26679417
- [Background] Jeng B, Cederberg KLJ, Lai B, Sasaki JE, Bamman MM, Motl RW. Oxygen cost of over-ground walking in persons with mild-to-moderate Parkinson's disease. Gait Posture. 2020 Oct;82:1-5. doi: 10.1016/j.gaitpost.2020.08.108. Epub 2020 Aug 11. PMID 32836026
- [Background] Kitada T, Pisani A, Porter DR, Yamaguchi H, Tscherter A, Martella G, Bonsi P, Zhang C, Pothos EN, Shen J. Impaired dopamine release and synaptic plasticity in the striatum of PINK1-deficient mice. Proc Natl Acad Sci U S A. 2007 Jul 3;104(27):11441-6. doi: 10.1073/pnas.0702717104. Epub 2007 Jun 11. PMID 17563363
- [Background] La Marca M, Beffy P, Pugliese A, Longo V. Fermented wheat powder induces the antioxidant and detoxifying system in primary rat hepatocytes. PLoS One. 2013 Dec 31;8(12):e83538. doi: 10.1371/journal.pone.0083538. eCollection 2013. PMID 24391783
- [Background] Lee MK, Stirling W, Xu Y, Xu X, Qui D, Mandir AS, Dawson TM, Copeland NG, Jenkins NA, Price DL. Human alpha-synuclein-harboring familial Parkinson's disease-linked Ala-53 --> Thr mutation causes neurodegenerative disease with alpha-synuclein aggregation in transgenic mice. Proc Natl Acad Sci U S A. 2002 Jun 25;99(13):8968-73. doi: 10.1073/pnas.132197599. PMID 12084935
- [Background] Liang J, Zhang XY, Zhen YF, Chen C, Tan H, Hu J, Tan MS. PGK1 depletion activates Nrf2 signaling to protect human osteoblasts from dexamethasone. Cell Death Dis. 2019 Nov 26;10(12):888. doi: 10.1038/s41419-019-2112-1. PMID 31767834
- [Background] Liu W, Wang C, He T, Su M, Lu Y, Zhang G, Munte TF, Jin L, Ye Z. Substantia Nigra Integrity Correlates with Sequential Working Memory in Parkinson's Disease. J Neurosci. 2021 Jul 21;41(29):6304-6313. doi: 10.1523/JNEUROSCI.0242-21.2021. PMID 34099507
- [Background] Ma Q. Role of nrf2 in oxidative stress and toxicity. Annu Rev Pharmacol Toxicol. 2013;53:401-26. doi: 10.1146/annurev-pharmtox-011112-140320. PMID 23294312
- [Background] Martella G, Madeo G, Maltese M, Vanni V, Puglisi F, Ferraro E, Schirinzi T, Valente EM, Bonanni L, Shen J, Mandolesi G, Mercuri NB, Bonsi P, Pisani A. Exposure to low-dose rotenone precipitates synaptic plasticity alterations in PINK1 heterozygous knockout mice. Neurobiol Dis. 2016 Jul;91:21-36. doi: 10.1016/j.nbd.2015.12.020. Epub 2016 Feb 23. PMID 26916954
- [Background] Padmanabhan P, Sreekanth Rao K, Gonzalez AJ, Pantelyat AY, Chib VS, Roemmich RT. The Cost of Gait Slowness: Can Persons with Parkinson's Disease Save Energy by Walking Faster? J Parkinsons Dis. 2021;11(4):2073-2084. doi: 10.3233/JPD-212613. PMID 34511512
- [Background] Petrillo S, Schirinzi T, Di Lazzaro G, D'Amico J, Colona VL, Bertini E, Pierantozzi M, Mari L, Mercuri NB, Piemonte F, Pisani A. Systemic activation of Nrf2 pathway in Parkinson's disease. Mov Disord. 2020 Jan;35(1):180-184. doi: 10.1002/mds.27878. Epub 2019 Nov 4. PMID 31682033
- [Background] Ponterio G, Tassone A, Sciamanna G, Vanni V, Meringolo M, Santoro M, Mercuri NB, Bonsi P, Pisani A. Enhanced mu opioid receptor-dependent opioidergic modulation of striatal cholinergic transmission in DYT1 dystonia. Mov Disord. 2018 Feb;33(2):310-320. doi: 10.1002/mds.27212. Epub 2017 Nov 18. PMID 29150865
- [Background] Rothman DL, Dienel GA, Behar KL, Hyder F, DiNuzzo M, Giove F, Mangia S. Glucose sparing by glycogenolysis (GSG) determines the relationship between brain metabolism and neurotransmission. J Cereb Blood Flow Metab. 2022 May;42(5):844-860. doi: 10.1177/0271678X211064399. Epub 2022 Jan 7. PMID 34994222
- [Background] Sciamanna G, Ponterio G, Vanni V, Laricchiuta D, Martella G, Bonsi P, Meringolo M, Tassone A, Mercuri NB, Pisani A. Optogenetic Activation of Striatopallidal Neurons Reveals Altered HCN Gating in DYT1 Dystonia. Cell Rep. 2020 May 19;31(7):107644. doi: 10.1016/j.celrep.2020.107644. PMID 32433955
- [Background] Spolaor F, Romanato M, Annamaria G, Peppe A, Bakdounes L, To DK, Volpe D, Sawacha Z. Relationship between Muscular Activity and Postural Control Changes after Proprioceptive Focal Stimulation (Equistasi(R)) in Middle-Moderate Parkinson's Disease Patients: An Explorative Study. Sensors (Basel). 2021 Jan 14;21(2):560. doi: 10.3390/s21020560. PMID 33466838
- [Background] Storm FA, Cesareo A, Reni G, Biffi E. Wearable Inertial Sensors to Assess Gait during the 6-Minute Walk Test: A Systematic Review. Sensors (Basel). 2020 May 6;20(9):2660. doi: 10.3390/s20092660. PMID 32384806
- [Background] Tassone A, Martella G, Meringolo M, Vanni V, Sciamanna G, Ponterio G, Imbriani P, Bonsi P, Pisani A. Vesicular Acetylcholine Transporter Alters Cholinergic Tone and Synaptic Plasticity in DYT1 Dystonia. Mov Disord. 2021 Dec;36(12):2768-2779. doi: 10.1002/mds.28698. Epub 2021 Jun 26. PMID 34173686
- [Background] Tyrrell DJ, Bharadwaj MS, Van Horn CG, Marsh AP, Nicklas BJ, Molina AJ. Blood-cell bioenergetics are associated with physical function and inflammation in overweight/obese older adults. Exp Gerontol. 2015 Oct;70:84-91. doi: 10.1016/j.exger.2015.07.015. Epub 2015 Jul 29. PMID 26226578
- [Background] Valdinocci D, Simoes RF, Kovarova J, Cunha-Oliveira T, Neuzil J, Pountney DL. Intracellular and Intercellular Mitochondrial Dynamics in Parkinson's Disease. Front Neurosci. 2019 Sep 18;13:930. doi: 10.3389/fnins.2019.00930. eCollection 2019. PMID 31619944
- [Background] Wang Y, Gao L, Chen J, Li Q, Huo L, Wang Y, Wang H, Du J. Pharmacological Modulation of Nrf2/HO-1 Signaling Pathway as a Therapeutic Target of Parkinson's Disease. Front Pharmacol. 2021 Nov 23;12:757161. doi: 10.3389/fphar.2021.757161. eCollection 2021. PMID 34887759
- [Background] Wertman V, Gromova A, La Spada AR, Cortes CJ. Low-Cost Gait Analysis for Behavioral Phenotyping of Mouse Models of Neuromuscular Disease. J Vis Exp. 2019 Jul 18;(149):10.3791/59878. doi: 10.3791/59878. PMID 31380846
- [Background] Zampese E, Surmeier DJ. Calcium, Bioenergetics, and Parkinson's Disease. Cells. 2020 Sep 8;9(9):2045. doi: 10.3390/cells9092045. PMID 32911641
- [Background] Zane AC, Reiter DA, Shardell M, Cameron D, Simonsick EM, Fishbein KW, Studenski SA, Spencer RG, Ferrucci L. Muscle strength mediates the relationship between mitochondrial energetics and walking performance. Aging Cell. 2017 Jun;16(3):461-468. doi: 10.1111/acel.12568. Epub 2017 Feb 9. PMID 28181388